CLINICAL TRIAL: NCT00659412
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Alefacept When Given in Combination With Methotrexate in Subjects With Psoriatic Arthritis With an Open-label Retreatment Course
Brief Title: A Placebo-controlled Study With an Extension Examining the Safety and Efficacy of Alefacept in Psoriatic Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-737
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic arthritis; psoriasis; Alefacept
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis | interventions — Alefacept; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Course A1 (Experimental)
  Interventions: Drug: Alefacept; Drug: Methotrexate
- Course A2 (Placebo Comparator)
  Interventions: Drug: Methotrexate; Drug: Placebo
- Course B (Experimental): Open-label extension
  Interventions: Drug: Alefacept; Drug: Methotrexate

INTERVENTIONS:
Drug: Alefacept — Intramuscular
  Other Names: Amevive, ASP0485
  Arms: Course A1; Course B
Drug: Methotrexate — Oral
Drug: Placebo — Intramuscular
  Arms: Course A2

SUMMARY:
Randomized, double-blind, 24-week study of patients with psoriatic arthritis comparing alefacept + methotrexate (MTX) vs. placebo + MTX followed by a 24-week open-label extension with only alefacept + MTX treatment.

DETAILED DESCRIPTION:
Patients who completed the initial 24-week treatment course and met the inclusion and exclusion criteria for the 24 week open-label extension continued on their stable MTX dose and also received alefacept throughout this extension.

ELIGIBILITY:
Inclusion Criteria:

* Psoriatic arthritis
* MTX treatment for 3 months prior to enrollment with continuing disease
* Normal T-cell count

Exclusion Criteria:

* Other types of psoriasis
* History of malignancy or lymphoproliferative disorder
* Serious infection or fever
* Antibody positive for Hepatitis C, HIV or TB
* Hepatic transaminases > 2X normal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2003-09; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving a score in the assessment system of the American College of Rheumatology Core Set Measurements of ACR 20, ACR 50 and ACR 70 | 12 Weeks and at any time

SECONDARY OUTCOMES:
Proportion of patients achieving a score in the Psoriasis Area and Severity Index of PASI 75, PASI 50 and PASI 25 | Each scheduled efficacy visit
Proportion of patients achieving a classification in the Physician's Global Assessment (PGA) of clear/almost clear | Each scheduled efficacy visit
Sharp -VanDen Heijde Modified Score of Joint Damage (X-ray) | Baseline, 24 Weeks and 48 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (24):
- United States (5):
  - Birmingham, Alabama
  - Wheaton, Maryland
  - Lake Success, New York
  - Rochester, New York
  - Seattle, Washington
- Canada (6):
  - Victoria, British Columbia
  - St. John's, Newfoundland and Labrador
  - London, Ontario
  - Newmarket, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Germany (3):
  - Berlin
  - Frankfurt
  - Göttingen
- Poland (6):
  - Bialystok
  - Elblag
  - Kalisz
  - Krakow
  - Torun
  - Warsaw
- Russia (4):
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Yaroslavl

REFERENCES:
- [Background] Mease PJ, Gladman DD, Keystone EC; Alefacept in Psoriatic Arthritis Study Group. Alefacept in combination with methotrexate for the treatment of psoriatic arthritis: results of a randomized, double-blind, placebo-controlled study. Arthritis Rheum. 2006 May;54(5):1638-45. doi: 10.1002/art.21870. PMID 16646026
- [Background] Mease PJ, Reich K; Alefacept in Psoriatic Arthritis Study Group. Alefacept with methotrexate for treatment of psoriatic arthritis: open-label extension of a randomized, double-blind, placebo-controlled study. J Am Acad Dermatol. 2009 Mar;60(3):402-11. doi: 10.1016/j.jaad.2008.09.050. Epub 2008 Nov 25. PMID 19028407